CLINICAL TRIAL: NCT04699721
Title: Clinical Study of Neoadjuvant Chemotherapy and Immunotherapy Combined With Probiotics in Patients With Resectable Non-small Cell Lung Cancer
Brief Title: Clinical Study of Neoadjuvant Chemotherapy and Immunotherapy Combined With Probiotics in Patients With Resectable NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202007093
Record Dates: First submitted 2020-12-27; First posted 2021-01-07 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-07

CONDITIONS: Non-small Cell Lung Cancer Stage II; Non-small Cell Lung Cancer Stage ⅢA; Non-small Cell Lung Cancer Stage IIIB
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Paclitaxel; Short Interspersed Nucleotide Elements

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): 3 cycles of nivolumab+Paclitaxel (albumin-bound type)+ Carboplatin AUC5 (21 days/cycle); as well as BiFico (oral taking, 4 capsules/time, 2 times per day)
  Interventions: Drug: nivolumab 4.5mg/kg+Paclitaxel (albumin-bound type) 260mg / m2+ Carboplatin AUC5

INTERVENTIONS:
Drug: nivolumab 4.5mg/kg+Paclitaxel (albumin-bound type) 260mg / m2+ Carboplatin AUC5 — 3 cycles of nivolumab+Paclitaxel (albumin-bound type)+ Carboplatin AUC5 (21 days/cycle); as well as BiFico (oral taking, 4 capsules/time, 2 times per day)
  Other Names: Bifidobacterium trifidum live powder (BiFico, SINE)

SUMMARY:
To evaluate the safety and effect of neoadjuvant chemotherapy and immunotherapy combined with probiotics for early resectable NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed previously untreated non-small cell lung cancer. Patients with stage II, IIIA and potentially resectable stage IIIB (T3N2) disease (according to AJCC 8th edition) are eligible ;
* Eastern Cooperative Oncology Group (ECOG) performance status score 0-1;
* 18 years ≤ Age ≤ 80 years. Signed and dated written informed consent must be provided by the patient prior to admission to the study;
* Patients with appropriate treatment compliance and could be followed-up correctly;
* Patients with measurable or evaluable diseases (according to RECIST 1.1);
* Patients must have the ability to swallow oral drugs;
* Patients with adequate pulmonary function capable of tolerating the proposed lung resection (as determined by the surgeon);
* Signed and dated written informed consent must be provided by the patient prior to admission to the study.

Exclusion Criteria:

* Subjects with known ALK translocations or EGFR mutations.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll;
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease;
* Patients with symptomatic ILD (grade 3-4) and/or poor lung function and a history of interstitial lung disease cannot be included. If you have any questions, please contact the trial team;
* Patients with other active malignant tumors currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug;
* Patients who are inability to follow the procedures required in the protocol due to any medical, mental or psychological conditions;
* Prior treatment with an anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibody or any other antibodies or drugs that target T cell costimulation or immune checkpoint pathways;
* Known positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid indicating acute or chronic infection;
* Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome;
* Patients with a history of allergy to study drugs or ingredients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | Within 3 days after the operation
  The percentage of participants with 0% residual viable tumor cells in the primary tumor and sampled lymph nodes after neoadjuvant therapy, as assessed by a blinded independent pathological review.

SECONDARY OUTCOMES:
Objective response rate | 28 days after the completion of three cycles of neoadjuvant therapy and before the operation
  The percentage of participants who achieved complete response or partial response after 3 cycles of neoadjuvant therapy according to the RECIST 1.1 criteria.
Major Pathologic Response | Within 3 days after the operation
  The percentage of participants with no more than 10% residual viable tumor cells in the primary tumor and sampled lymph nodes after neoadjuvant therapy, as assessed by a blinded independent pathological review.
Disease free survival | 1 year, 3 years and 5 years after the operation
  The time (month) from the completion of lung cancer radical surgery to the recurrence or metastasis of the disease.
Recurrence rate | 1 year, 3 years and 5 years after the operation
  The percentage of participants who have recurrence or metastasis of lung cancer at certain time points after radical surgery.
Overall survival | 1 year, 3 years and 5 years after the operation
  The time (month) from the completion of lung cancer radical surgery to all-cause death.
Adverse effects | Treatment-related adverse events were assessed between the first neoadjuvant dose and 30 days after the last dose of neoadjuvant study treatment.
  The number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Surgical complications (intra-operative and peri-operative) | 90 days after the first medication or 30 days after the operation, whichever is later
  The number of participants with surgery-related adverse events that occur during or after a surgical procedure.
R0 surgical events | 28 days after the completion of three cycles of neoadjuvant therapy
  The number of participants who have lung cancer completely resected. It is defined as the removal of negative margins, encompassing bronchial, arterial, venous peribronchial, and surrounding tissues near the tumor. In addition, at least 6 groups of lymph nodes must be removed, including at least 3 groups of intrapulmonary lymph nodes and 3 groups of mediastinal lymph nodes (station 7 lymph node must be included). The resected lymph nodes should be negative upon microscopic examination.
Clinical TNM downstaging | 28 days after the completion of three cycles of neoadjuvant therapy and before the operation
  The number of participants who achieve a decrease in the clinical TNM stage of lung cancer following neoadjuvant therapy before surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Gao, Doctor, Study Director — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: IPD will be shared when the clinical trail is finished